CLINICAL TRIAL: NCT04912544
Title: Feasibility and Intelligibility Testing of a Microphone System to Facilitate Patient Communication During Noninvasive Ventilation
Brief Title: Facilitating Patient Communication During Noninvasive Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Axon Medical, Inc. (Unknown); Intermountain Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sarah Ferguson, Associate Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 00056030; 1R43HL147788-01A1 (NIH)
Record Dates: First submitted 2021-04-28; First posted 2021-06-03 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Noninvasive Ventilation; Speech Intelligibility
MeSH Terms: conditions — Speech Intelligibility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Patient talking with microphone first turned on and then off
  Interventions: Device: Noninvasive Ventilation Mask Microphone
- Arm 2 (Experimental): Patient talking with microphone first turned off and then on
  Interventions: Device: Noninvasive Ventilation Mask Microphone

INTERVENTIONS:
Device: Noninvasive Ventilation Mask Microphone — Noninvasive Ventilation Mask Microphone is turned on to enhance speech intelligibility during the intervention portion of the crossover feasibility study

SUMMARY:
Assessing speech intelligibility in a pilot study of patients speaking with a mask microphone while being treated with standard of care non-invasive ventilation. This is a feasibility study to test the microphone in a real world setting.

DETAILED DESCRIPTION:
We will conduct a prospective feasibility study to evaluate speech intelligibility of 10 patients (target distribution of gender: 5 males, 5 females) undergoing standard of care, clinically indicated non-invasive ventilation. Patients will be their own control with and without the ReddyPort™ microphone using a crossover design, with the sequence of conditions randomized (half of patients start with microphone turned on, half start with the microphone turned off). The patients in this study will all receive standard of care. No medical decisions for a change in care will result from the speech recordings obtained during this feasibility study. The speech recordings will be analyzed off-site using a pool of blinded volunteers. The microphone on and off test conditions will not be used to change outcome of the clinical course of care.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Currently hospitalized
* Awake and able to attempt communication
* Respiratory failure requiring non-invasive ventilatory support
* Positive Inspiratory Pressure (PIP) less than or equal to 20 cm H2O
* Positive End Expiratory Pressure (PEEP) less than or equal to 10 cm H2O
* FiO2 less than or equal to 0.60
* Clinical attending physician believes it is safe for the patient to participate
* Able to consent o If patient cannot consent on the basis of difficulty in being heard and asking questions (as in fact may occur with NIV, a key assumption of this study), then assent will be obtained from the patient with informed consent obtained from a legally authorized representative.

Exclusion Criteria:

* Tachypnea with RR > 35
* Increase in PIP, PEEP or FiO2 over the last 2 hours
* Known to be delirious (clinically obtained CAM score that is positive)
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Rating of speech intelligibility | Intelligibility will be rated offline by blinded listeners who hear the recording 1-12 weeks after speaking tasks are complete.
  The 1-5 likert scale developed by Yorkston et al will be used to evaluate speech intelligibility of the device (Yorkston, Kathryn M., David R. Beukelman, and Charles Traynor. Assessment of intelligibility of dysarthric speech. Austin, TX: Pro-ed, 1984.Powell TW. A comparison of English reading passages for elicitation of speech samples from clinical populations. Clin Linguist Phon. 2006;20(2-3):91-7)

SECONDARY OUTCOMES:
Rating of microphone likability | Immediately after speaking tasks are complete
  Subjects will be asked how well they liked using the microphone on a Likert-type scale of 1-5, from extremely unlikable (1) to extremely likable (5)
Rating of speech comprehensibility | Immediately after speaking tasks are complete
  Subjects will be asked how well they could understand the speech on a Likert-type scale of 1-5, from not at all understandable (1) to fully understandable (5)
Rating of how natural the speech sound quality is | Immediately after speaking tasks are complete
  Subjects will be asked how natural the speech sound quality is on a Likert-type scale of 1-5, from not natural (1) to completely natural (5)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Brewer, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No